CLINICAL TRIAL: NCT00782340
Title: Phase III, Multi-Center, Study to Assess the Clinical Effect of Droxidopa in Subjects With Primary Autonomic Failure, Dopamine Beta Hydroxylase Deficiency or Non-Diabetic Neuropathy and Symptomatic NOH
Brief Title: A Clinical Study for Patients With Neurogenic Orthostatic Hypotension (NOH) Using Droxidopa
Acronym: NOH301
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chelsea Therapeutics (Industry)
Collaborators: Chiltern International Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Droxidopa NOH301; NCT00879567 (obsolete NCT alias)
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2014-05-16 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: Symptomatic Neurogenic Orthostatic Hypotension (NOH); Non-diabetic Neuropathy; Primary Autonomic Failure; Dopamine Beta Hydroxylase Deficiency
Keywords: NOH; Neurogenic Orthostatic Hypotension; Orthostatic hypotension; PAF; Pure Autonomic Failure; MSA; Multiple System Atrophy; Neuropathy; Autonomic Failure; Parkinson; Dopamine Deficiency; Dopamine; Droxidopa
MeSH Terms: conditions — dopamine beta hydroxylase deficiency; Hypotension, Orthostatic; Pure Autonomic Failure; Multiple System Atrophy | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Droxidopa (Active Comparator): 100 mg, oral, three times per day 200 mg, oral, three times per day 300 mg, oral, three times per day 400 mg, oral, three times per day 500 mg, oral, three times per day 600 mg, oral, three times per day
  Interventions: Drug: Droxidopa
- Placebo (Placebo Comparator): 100 mg, oral, three times per day 200 mg, oral, three times per day 300 mg, oral, three times per day 400 mg, oral, three times per day 500 mg, oral, three times per day 600 mg, oral, three times per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 100 mg, oral, three times per day 200 mg, oral, three times per day 300 mg, oral, three times per day 400 mg, oral, three times per day 500 mg, oral, three times per day 600 mg, oral, three times per day
  Arms: Placebo
Drug: Droxidopa — 100 mg, oral, three times per day 200 mg, oral, three times per day 300 mg, oral, three times per day 400 mg, oral, three times per day 500 mg, oral, three times per day 600 mg, oral, three times per day
  Arms: Droxidopa

SUMMARY:
The purpose of this study is to see whether droxidopa is effective in treating symptoms of neurogenic orthostatic hypotension in patients with Primary Autonomic Failure (Pure Autonomic Failure, Multiple System Atrophy, Parkinson's Disease), Non-diabetic neuropathy, or Beta Hydroxylase deficiency.

DETAILED DESCRIPTION:
Systolic blood pressure is transiently and minimally decreased in healthy individuals upon standing. Normal physiologic feedback mechanisms work through neurally-mediated pathways to maintain the standing blood pressure, and thus maintain adequate cerebral perfusion. The compensatory mechanisms that regulate blood pressure upon standing are dysfunctional in subjects with orthostatic hypotension (OH), a condition that may lead to inadequate cerebral perfusion with accompanying symptoms of syncope, dizziness or lightheadedness, unsteadiness and blurred or impaired vision, among other symptoms.

The autonomic nervous system has a central role in the regulation of blood pressure. Primary Autonomic Failure is manifested in a variety of syndromes. Orthostatic hypotension is a usual presenting symptom. Primary Autonomic Failure may be the primary diagnosis, and classifications include pure autonomic failure (PAF), also called idiopathic orthostatic hypotension (Bradbury-Eggleston syndrome) autonomic failure with multiple system atrophy (Shy-Drager syndrome) and also Parkinson's disease. Regardless of the primary condition, autonomic dysfunction underlies orthostatic hypotension.

Orthostatic hypotension may be a severely disabling condition which can seriously interfere with the quality of life of afflicted subjects. Currently available therapeutic options provide some symptomatic relief in a subset of subjects, but are relatively ineffective and are often accompanied by severe side effects that limit their usefulness. Support garments (tight-fitting leotard) may prove useful in some subjects, but is difficult to don without family or nursing assistance, especially for older subjects. Midodrine, fludrocortisone, methylphenidate, ephedrine, indomethacin and dihydroergotamine are among some of the pharmacological interventions that have been used to treat orthostatic hypotension, although only midodrine is specifically approved for this indication. The limitations of these currently available therapeutic options, and the incapacitating nature and often progressive downhill course of disease, point to the need for an improved therapeutic alternative.

The current withdrawal design study will measure the efficacy of droxidopa on symptoms of neurogenic orthostatic hypotension in patients randomized to continued droxidopa treatment versus placebo, following 14 days of double-blind treatment.

droxidopa

droxidopa [also, known as L-threo-3,4-dihydroxyphenylserine, L-threo-DOPS, or L-DOPS] is the International non-proprietary name (INN) for a synthetic amino acid precursor of norepinephrine (NE), which was originally developed by Sumitomo Pharmaceuticals Co., Limited, Japan. It has been approved for use in Japan since 1989. Droxidopa has been shown to improve symptoms of orthostatic hypotension that result from a variety of conditions including Shy Drager syndrome (Multiple System Atrophy), Pure Autonomic Failure, and Parkinson's disease. There are four stereoisomers of DOPS; however, only the L-threo-enantiomer (droxidopa) is biologically active.

The exact mechanism of action of droxidopa in the treatment of symptomatic NOH has not been precisely defined; however, its NE replenishing properties with concomitant recovery of decreased noradrenergic activity are considered to be of major importance.

Droxidopa has been marketed in Japan since 1989. Data from clinical studies and post-marketing surveillance programs conducted in Japan show that the most commonly reported adverse drug reactions with droxidopa are increased blood pressure, nausea, and headache. In clinical studies, the prevalence and severity of droxidopa adverse effects appear to be similar to those reported by the placebo control arm.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, each patient must fulfill the following criteria:

* Male or female and aged 18 years or over
* Clinical diagnosis of orthostatic hypotension associated with Primary Autonomic Failure (PD, MSA and PAF), Dopamine Beta Hydroxylase Deficiency or Non-Diabetic Autonomic Neuropathies
* A documented fall in systolic blood pressure of at least 20 mmHg, or in diastolic blood pressure of at least 10 mmHg, within 3 minutes after standing;
* Provide written informed consent to participate in the study and understand that they may withdraw their consent at any time without prejudice to their future medical care.

Exclusion Criteria:

* Currently taking ephedrine or midodrine
* Patients taking ephedrine or midodrine must stop taking these drugs at least 2 days prior to their baseline visit (Visit 2).
* The use of short-acting anti-hypertensive medications at bedtime is permitted.
* Currently taking tri-cyclic antidepressant medication or other norepinephrine re-uptake inhibitors;
* Have changed dose, frequency and or type of prescribed medication, within two weeks of study start (excluding ephedrine and midodrine)
* History of more than moderate alcohol consumption
* History of known or suspected drug or substance abuse
* Women of childbearing potential who are not using a medically accepted contraception
* For WOCP a serum beta HCG pregnancy test must be conducted at screening, and a urine pregnancy test must be conducted at baseline and study termination; the results must be negative at screening and at baseline for the patient to receive study medication.
* Sexually active males whose partner is a WOCP and who do not agree to use condoms for the duration of the study and for 30 days after the last dose;
* Women who are pregnant or breast feeding
* Known or suspected hypersensitivity to the study medication or any of its ingredients
* Pre-existing sustained severe hypertension (BP 180/110 mmHg in the sitting position)
* Have atrial fibrillation or, in the investigator's opinion, have any other significant cardiac arrhythmia
* Any other significant systemic, hepatic, cardiac or renal illness
* Diabetes mellitus or insipidus
* Have a history of closed angle glaucoma
* Have a known or suspected malignancy
* Have a serum creatinine level > 130 mmol/L
* Patients with known gastrointestinal illness or other gastrointestinal disorder that may, in the investigator's opinion, affect the absorption of study drug
* In the investigator's opinion, have clinically significant abnormalities on clinical examination or laboratory testing
* In the investigator's opinion, are unable to adequately co-operate because of individual or family situation
* In the investigator's opinion, are suffering from a mental disorder that interferes with the diagnosis and/or with the conduct of the study, e.g. schizophrenia, major depression, dementia
* Are not able or willing to comply with the study requirements for the duration of the study
* Have participated in another clinical trial with an investigational agent (including named patient or compassionate use protocol) within 4 weeks before the start of the study
* Previous enrolment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Greer, MD, Principal Investigator — Arkansas Cardiology; Alberto Vasquez, MD, Principal Investigator — Suncoast Neuroscience; Richard Hull, MD, Principal Investigator — North Alabama Neuroscience; Brent Goodman, MD, Principal Investigator — Mayo Clinic; Alvin McElveen, MD, Principal Investigator — Bradenton Neurology, Inc; Mazen Dimachkie, MD, Principal Investigator — University of Kansas Medical Center
Locations (21):
- United States (14):
  - North Alabama Neuroscience, Huntsville, Alabama
  - Mayo Clinic-Arizona, Scottsdale, Arizona
  - Arkansas Cardiology, Little Rock, Arkansas
  - University of California, Irvine, Irvine, California
  - Bradenton Neurology, Inc, Bradenton, Florida
  - Suncoast Neuroscience Associates, Inc, St. Petersburg, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cncs, Ninds,Nih, Bethesda, Maryland
  - Nerological Reserch Center at Hattiesburg, Hattiesburg, Mississippi
  - North Shore Hospital, Manshasette, New York
  - Pennsylvania Hospital of the University of PA Health System- Department of Neurology, Philadelphia, Pennsylvania
  - HAN Neurological Associates, Upland, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Evergreen Hospital Medical Center; Booth Gardner Parkinson's Care Center, Kirkland, Washington
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Movment Disorder Clinic Deer lodge Centre, Winnipeg, Manitoba
  - David B. King, - Private Clinic, Halifax, Nova Scotia
  - London Health Sciences Centre, UH, London, Ontario
  - UHNresearch, Toronto, Ontario
  - IRCM, Montreal, Quebec

REFERENCES:
- [Derived] Biaggioni I, Arthur Hewitt L, Rowse GJ, Kaufmann H. Integrated analysis of droxidopa trials for neurogenic orthostatic hypotension. BMC Neurol. 2017 May 12;17(1):90. doi: 10.1186/s12883-017-0867-5. PMID 28494751
- [Derived] Francois C, Rowse GJ, Hewitt LA, Vo P, Hauser RA. Analysis of number needed to treat for droxidopa in patients with symptomatic neurogenic orthostatic hypotension. BMC Neurol. 2016 Aug 18;16(1):143. doi: 10.1186/s12883-016-0665-5. PMID 27538531

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Label Titration: All patients titrated to their optimal dose of droxidopa for up to 2 weeks during open-label dose titration.
Period: Open Label Titration
Arm/Group | Open-Label Titration | Droxidopa | Placebo
Started | 263 | 0 | 0
Completed | 162 | 0 | 0
Not Completed | 101 | 0 | 0
Not completed — Adverse Event | 12 | 0 | 0
Not completed — Treatment failure | 50 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0
Not completed — Enrollment capped | 16 | 0 | 0
Not completed — Did not meet responder criteria | 2 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0
Not completed — Randomized in error | 6 | 0 | 0
Period: Randomized Double Blind
Arm/Group | Open-Label Titration | Droxidopa | Placebo
Started | 0 | 82 | 80
Completed | 0 | 82 | 80
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Not Randomized: Patients entered open label droxidopa dose titration, but did not proceed into washout and randomization.
- Total: Total of all reporting groups
Arm/Group | Not Randomized | Droxidopa | Placebo | Total
Number analyzed (Participants) | 101 | 82 | 80 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (15.4) | 57.4 (16.90) | 55.7 (20.03) | 59.6 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 40 | 38 | 115
  Male | 64 | 42 | 42 | 148
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 99 | 82 | 78 | 259
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 48 | 33 | 32 | 113
  Canada | 3 | 0 | 4 | 7
  Europe | 50 | 49 | 44 | 143
Primary Clinical Diagnosis [Number; unit: participants]
  Parkinson's Disease | 45 | 35 | 31 | 111
  Multiple System Atrophy | 18 | 15 | 11 | 44
  Pure Autonomic Failure | 33 | 26 | 28 | 87
  Non-Diabetic Autonomic Neuropathy | 2 | 2 | 6 | 10
  Other Diagnosis | 3 | 4 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Orthostatic Hypotension Questionnaire Score (OHQ)
Description: The OHQ is the average of two sub-scales, the Orthostatic Hypotension Symptom Assessment Scale (OHSA) and the Orthostatic Hypotension Daily Activities Scale (OHDAS). Each asks the patient to rate their symptoms or disease impact over the past week. The OHSA sub-scale is the average of six items: 1) Dizziness, lightheadedness, feeling faint or feeling like you might black out; 2) Problems with vision; 3) Weakness; 4) Fatigue; 5) Trouble concentrating; and 6) Head/neck discomfort. The OHDAS sub-scale is the average of four items: 1) Standing for a short time; 2) Standing for a long time; 3) Walking for a short time; and 4) Walking for a long time. Each item is scored on a Likert scale from 0 to 10, with 10 being the most severe.
  For the change from randomization, negative numbers represent improvement from randomization in OHQ score.
Time Frame: 7 days
Population: Missing data are imputed using the last observation carried forward method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 82 | 80
units on a scale | -1.83 (2.067) | -0.93 (1.691)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — Statistical analysis plan involved a hierarchical assessment of secondary endpoints to prevent inflation of type I errors; ANCOVA model that includes treatment as a factor and baseline OHQ composite score as a co-variate

2. Secondary Outcome: Change in Ability to Conduct Activities of Daily Living Score (OHDAS Composite Score)
Description: OHDAS composite scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. A negative score indicates an improvement during the double-blind randomized phase relative to value at randomization.
Time Frame: 7 days
Population: Missing data are imputed using the last observation carried forward method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 81 | 79
units on a scale | -1.98 (2.310) | -0.92 (1.816)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model that includes treatment as a factor and baseline OHDAS composite score as a co-variate

3. Secondary Outcome: Change in Orthostatic Hypotension Symptom Assessment (OHSA Composite) Score
Description: OHSA composite scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. A negative score indicates an improvement during the double-blind randomized phase relative to value at randomization.
Time Frame: 7 days
Population: Missing data are imputed using the last observation carried forward method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 81 | 79
units on a scale | -1.68 (2.125) | -0.95 (1.901)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.010, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model including a factor for randomized treatment along with the OHSA composite value at randomization as a covariate

4. Secondary Outcome: Change in Activities Involving Standing a Short Time (OHDAS Item 1)
Description: OHDAS Item 1 scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. A negative score indicates an improvement during the double-blind randomized phase relative to value at randomization.
Time Frame: 7 days
Population: Missing data are imputed using the last observation carried forward method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 82 | 80
units on a scale | -1.9 (2.75) | -0.8 (2.60)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.003, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; Mantel-Haenszel statistic comparing treatment groups based on rank statistics adjusted for the covariate OHSA Item 1 value at baseline

5. Secondary Outcome: Change in Activities Involving Walking a Short Time (OHDAS Item 3)
Description: OHDAS Item 3 scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. A negative score indicates an improvement during the double-blind randomized phase relative to value at randomization.
Time Frame: 7 days
Population: Missing data are imputed using the last observation carried forward method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 82 | 80
units on a scale | -1.7 (2.55) | -0.6 (2.37)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.009, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 3, analysis 1]

6. Secondary Outcome: Change in Dizziness/ Lightheadedness/ Feeling Faint/ or Feeling Like You Might Blackout (OHSA Item 1)
Description: OHSA item 1 scale range: 0 (none) -10 (worst), likert scale. Change: score at end of study minus score at randomization. A negative score indicates an improvement during the double-blind randomized phase relative to value at randomization.
Time Frame: 7 days
Population: Missing data are imputed using the last observation carried forward method.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 82 | 80
units on a scale | -2.4 (3.20) | -1.1 (2.58)
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p < 0.001, Mantel Haenszel — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 4, analysis 1]

7. Secondary Outcome: Patient-Reported Clinical Global Improvement - Severity Scores
Description: The CGI-S is a 7 point scale ranging from a score of 1 (no symptoms) to 7 (severe symptoms). Patients were grouped according to OH severity at the end of the randomization period as follows;
  Normal-Borderline OH (CGI-S 1-2), Mild-Moderate OH (CGI-S 3-4), Marked OH-Most Ill with OH (CGI-S 5-7).
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 82 | 80
participants
  Normal-Borderline OH | 23 | 16
  Mild-Moderate OH | 39 | 47
  Marked OH-Most ill with OH | 20 | 17
Statistical Analysis 1: Comparison: Droxidopa vs Placebo; Test type: Superiority or Other; p = 0.327, Fisher Exact — Statistical analysis plan involved a hierarchical assessment of secondary endpoints to prevent inflation of type I errors. As the this endpoint was not positive, no additional statistical analyses will be performed on secondary endpoints

8. Secondary Outcome: Clinician-Reported Clinical Global Improvement - Severity Scores
Description: as for outcome 7
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 82 | 80
participants
  Normal-Borderline OH | 21 | 15
  Mild-Moderate OH | 39 | 44
  Marked OH-Most ill with OH | 22 | 21

9. Secondary Outcome: Change in Systolic Blood Pressure (SBP) Measurements 3 Minutes Post Standing
Description: Change: standing systolic blood pressure at end of study minus standing systolic blood pressure at randomization. A positive score indicates an improvement during the double-blind randomized phase relative to value at randomization.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Droxidopa | Placebo
Number analyzed (Participants) | 82 | 79
mmHg | 11.2 (22.89) | 3.9 (16.28)

ADVERSE EVENTS:
Description: One patient randomized to the droxidopa group in the randomized double blind phase was treated with placebo during this period and is included in the placebo group (actual treatment received) for the safety analyses.
Groups:
- Open-Label Titration: All patients treated with study drug during dose titration (7-14 days)
Arm/Group | Open-Label Titration | Droxidopa | Placebo
Serious Adverse Events (participants affected / at risk) | 2/263 | 0/81 | 0/81
Other Adverse Events (participants affected / at risk) | 38/263 | 9/81 | 1/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Titration (N=263) | Droxidopa (N=81) | Placebo (N=81)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Titration (N=263) | Droxidopa (N=81) | Placebo (N=81)
Headache (Nervous system disorders) | 26 (34) | 6 (7) | 0 (0)
Dizziness (Nervous system disorders) | 17 (18) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less